CLINICAL TRIAL: NCT04526522
Title: Does Low Social Acceptance Among Peers Increase the Risk of Future Persistent Musculoskeletal Pain in Adolescents? Prospective Data From the Fit Futures Study
Brief Title: "Social Acceptance Among Peers and Musculoskeletal Pain in Adolescents"
Status: Completed | Type: Observational
Sponsor: Oslo Metropolitan University (Other)
Responsible Party: Principal Investigator, Britt Elin Øiestad, Associated Professor, Oslo Metropolitan University
Other Study IDs: 2019/599
Record Dates: First submitted 2019-12-19; First posted 2020-08-26 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Musculoskeletal Pain
Keywords: musculoskeletal pain; adolescent; risk factor
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Musculoskeletal pain is common and often occurs already in adolescence. To be able to target future interventions that aim to prevent new episodes of MSK pain, more studies on modifiable risk factors are necessary. In this prospective cohort study, already collected data from the Fit Futures study will be used. The aim is to investigate if perceived social acceptance among peers in the first year of high school is associated with musculoskeletal pain in the last year of high school, and if this association is moderated by psychological distress.

DETAILED DESCRIPTION:
Few studies have investigated social factors in association with musculoskeletal pain in adolescents, such as perceived peer acceptance. Adolescence is a vulnerable period of life when peer relations is important in order to develop social, emotional and behavioural skills. Social relations have been linked to several health outcomes in previous studies. Therefore, this study aims to investigate if social acceptance among peers is associated with musculoskeletal pain in adolescents.

The research questions are:

1. Is there a significant association between perceived social acceptance among peers during the first year of high school and persistent MSK pain two years later in adolescents?
2. Is psychological distress an effect modifier of the relationship between perceived social acceptance among peers during the first year of high school and MSK pain two years later in adolescents?

Method:

This is a prospective cohort study using data from the Fit Futures (FF) study. Students from the first year of high school were included at baseline in Fit Futures 1 (FF1) and followed up for two years later in Fit Futures 2 (FF2). The students answered a comprehensive questionnaire, including biological, psychological, and social variables. They also underwent measurements of height and weight during school hours.

Baseline characteristics will be extracted from FF1 with data collected in the period 2010-2011. Baseline characteristics from adolescents who participated in the study and adolescents who were lost to follow-up will be presented and compared. Information about age, sex, parents socioeconomic status (SES), and body mass index (BMI), will be used to describe the study sample and as potential confounders.

Social acceptance among peers was measured by five questions from the revised Norwegian version of Self-perception Profile for Adolescent; scale for social competence and psychological distress was measured by the Hopkins Symptoms Checklist-10.

Statistical analyses:

All statistical tests will be two-sided, and the nominal p-values will be reported. All confidence intervals (CIs) will be reported as 95%. Preliminary analyses of frequencies, missing data and normality will be conducted. The assumption of normal distribution will be investigated using histograms and QQ-plots. Normally distributed data will be described with means and standard deviations (SDs), skewed data will be presented with medians and ranges. Categorical data will be reported as counts and percentages. All statistical analyses will be conducted using SPSS statistical software (SPSS Inc, Chicago, IL, USA).

Participants with missing data on the outcome will be excluded from the analyses. Missing data on the exposure variable will be handled by multiple imputations unless the missingness is very low (<10%). A two-year incidence rate of participants who reports no MSK pain at baseline and develops persistent MSK pain during the follow-up period will be calculated, presented as percentage with 95% CI.

Logistic regression:

Main analyses will be conducted in a sample of adolescents that report no persistent MSK pain at baseline. Secondary analyses will be conducted in the total sample regardless of pain status at baseline. Binary logistic regression will be conducted with social acceptance among peers as the exposure and persistent MSK pain as the outcome. Sex and chronic diseases will be included as confounders.

Moderation analyses:

The moderation analysis will be performed as described by Hayes, using PROCESS macro model 1 in SPSS. In the analysis, social acceptance will be included as the exposure, MSK pain as the outcome, and psychological distress as the possible effect modifier. Sex and chronic diseases will be included as confounders. Regression coefficients and ORs will be presented in figures and tables. Confidence intervals for the effect modifier will be constructed using a bias-corrected bootstrap method with 5000 bootstrap samples.

Additional analyses:

Drop-out analyses will be conducted to explore possible attrition bias by comparing baseline characteristics between participants lost to follow-up and responders at follow-up. The chi-square test will be used for comparison of categorical variables, independent samples t-test to compare normally distributed continuous variables, and Mann-Whitney U test to compare data with skewed distribution.

ELIGIBILITY:
Inclusion criteria:

* Adolescents between 15 and 16 years who live in Tromsø or Balsfjord Municipality

Exclusion criteria (main analysis):

* Persistent MSK pain at baseline

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Norwegian adolescents of 15-18 years of age.
Sampling Method: Probability Sample
Enrollment: 961 (Actual)
Dates: Start 2010-09-01 (Actual); Primary Completion 2013-06-01 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Weekly musculoskeletal pain lasting for at least 3 months or more | 2 years
  Persistent or recurrent musculoskeletal pain lasting for at least 3 months or more. The questionnaire included question about pain duration in 14 body regions. Shoulder, arm/elbow, hand, hips, thigh/knee/shin, ankle, neck, upper back, lower back were used to define MSK pain based on the body regions from the Nordic Musculoskeletal Pain Questionnaire. The responses were yes or no, and duration ranged from everyday to rarer than every week.

SECONDARY OUTCOMES:
Severe weekly MSK pain lasting for at least 3 months or more | 2 years
  Persistent or recurrent MSK pain lasting for at least 3 months or more with a severity of at least 5 on a scale from 0-10 (0= no pain, 10=Worst pain imaginable). The questionnaire included question about pain duration in 14 body regions. Shoulder, arm/elbow, hand, hips, thigh/knee/shin, ankle, neck, upper back, lower back were used to define MSK pain based on the body regions from the Nordic Musculoskeletal Pain Questionnaire. The responses were yes or no, and duration ranged from everyday to rarer than every week.

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo Metropolitan University, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jahre H, Grotle M, Smedbraten K, Richardsen KR, Cote P, Steingrimsdottir OA, Nielsen C, Storheim K, Smastuen M, Stensland SO, Oiestad BE. Low social acceptance among peers increases the risk of persistent musculoskeletal pain in adolescents. Prospective data from the Fit Futures Study. BMC Musculoskelet Disord. 2022 Jan 13;23(1):44. doi: 10.1186/s12891-022-04995-6. PMID 35027018